CLINICAL TRIAL: NCT02487849
Title: Feasability of an Unique Intraoperative Given Hyperthermal Intraperitoneal Chemotherapy With Carboplatin During a Secondary Cytoreductive Operation in Patients With Platinum-sensitive Recurrence of Ovarian Carcinoma
Brief Title: HIPEC After Secondary Cytoreductive Operation in Patients With Platinum-sensitive Recurrence of Ovarian Carcinoma
Acronym: HIPEC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: actually limited personnel ressources
Sponsor: Krankenhaus Barmherzige Schwestern Linz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIPEC-OVAR-REZIDIV-2014-1.1; 2015-002436-41 (EudraCT Number)
Record Dates: First submitted 2015-06-13; First posted 2015-07-02 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Epithelial Ovarian Cancer; Peritoneal Cancer; Fallopian Tube Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms | interventions — Hyperthermic Intraperitoneal Chemotherapy; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HIPEC (Experimental): If patient is eligible - secondary cytoreductive operation will be followed by HIPEC with 800 mg/m² body surface (KOF) Carboplatin with closed technique.
  Interventions: Procedure: HIPEC; Drug: Carboplatin

INTERVENTIONS:
Procedure: HIPEC — secondary cytoreductive operation
  Other Names: Hyperthermal intraperitoneal Chemotherapy
Drug: Carboplatin — Hyperthermal Intraperitoneal Chemotherapy (HIPEC)
  Other Names: Carboplatin Accord

SUMMARY:
The combination of optimal cytoreductive operation (according to Desktop II criteria), HIPEC with Carboplatin 800 mg/m² KOF (Körperoberfläche) and following platinum-based systemic chemotherapy should be executed In patients with platinum-sensitive recurrence of ovarian carcinoma. Condition for HIPEC is attainment of optimal cytoreduction (R0) and experts judgement of a complication-free prolongation of narcosis after finishing the surgery. HIPEC will be administered additionally to standard therapy. If HIPEC was executed the number of systemic given platinum-based chemotherapy decreases for one cycle.

This regime should be investigated in terms of safety of performance, quality of life for the patients and consequences for the following systemic chemotherapy.

DETAILED DESCRIPTION:
In occurence with a platinum-sensitive recurrence of EOC survival can be prolonged by a recurrence-operation, if macroscopical tumor-free status (optimal cytoreductive operation) can be reached in combination with a platinum-based standard-chemotherapy.

Several studies showed that the combination of optimal cytoreductive operation and HIPEC is a secure method of treatment. In comparison to operation and standard-chemotherapy it has a significant positive influence on survival rates. A hyperthermal intraperitoneal chemotherapy with Carboplatin is possible without severe side-effects.

The combination of optimal cytoreductive operation (according to Desktop II criteria), HIPEC with Carboplatin and following platinum-based systemic chemotherapy should be carried out in patients with platinum-sensitive recurrence.

Condition for applying HIPEC is reaching optimal cytoreduction (<0.5 cm visible tumour rest at the end of operation) and according to expert opinion a complicatin-free prolongation of narcosis after finishing the operative intervention. HIPEC is carried out additionally to standard therapy. If it can be carried out, the amount of systemically administered patinum-based chemotherapy is reduced for one cycle.

This regime should be tested on safety in performance, quality of life for patients, and consequences for the following systemic chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years
* Signed informed consent
* Patients with platinum-sensitive recurrence after 12-48 months after platinum-based firstline-chemotherapy of histological saved epithelial ovarian carcinoma, primary peritoneal carcinoma or tube carcinoma with planned cytoreductive operation
* The following histological types can be included: serous, endometrioide, clear cell or undifferentiated carcinoma. Mixed epithelial carcinoma, malignant Brenner Tumour
* No preceding recurrence chemotherapy
* Preceding hormontherapy admitted. Concomitant antineoplastic antihormone-therapy (Tamoxifen, Aromataseinhibitoren etc.) not admitted. Low dosed (physiological) hormone-replacement-therapie (HRT) can be administered
* Patients with maintenance therapy (e.g. Bevacizumab) permitted, assumed recurrence was diagnosed 12 months after primary cytotoxic chemotherapy (also with maintenancetherapy during chemotherapy) and last administration of maintenancetherapy happened min. 21 days before first study protocol intervention
* Resectability R0 probably, fixed by Desktop II-criteria:
* Cytoreductive operation at first-diagnosis of the carcinoma R0
* Ascites <500 ml
* ECOG 0
* R0 status (≤0,5 cm tumour rest) at the end of secondary cytoreductive operation
* Eligibility for Standard systemic platinum-based combination chemotherapy after sec. cytoreductive operation with or without HIPEC (investigators decision)
* Bone marrow function: Haemoglobine ≥8.5 g/dL, Absol. neutrophile Granulocytes(ANC) ≥1.000/mm3, Thrombocytes ≥ 100.000/mm3
* Renal function: Serum Creatinin ≤1,5 times the ULN, calculated Creatininclearance (GFR) ≥60ml/min
* Liver function: Bilirubin ≤1,5 x
* ALT, AST ≤3 x ULN
* Adequate coagulation parameter: INR-value ≤1,5, aPTT ≤1,5 x ULN
* For patients under fully-dosed/therapeutic Warfarin- or Phenprocoumontherapy INR between 2-3 and aPTT <1,2 x ULN
* Neurol. Function: peripheral Neuropathy ≤Grade 2 (CTCAE v4.03 criteria)
* In women with childbearing potential availability of a neg. serum pregnancy test 2 weeks before planned sec. cytored. operation + effective contraception during study period guaranteed

Exclusion Criteria:

* No signed informed consent
* Tumours with low malignant potential (Borderline-carzinomas)
* Patients with preceding radiotherapy in abdomen and pelvis
* Patients with preceding endometrial carcinoma will be excluded, except: Stage IA [no low differentiated subtype (serous-papillary, clear cellular, FIGO grade 3)]
* With the exception of non-melanoma skin cancer and other specific malignancies as noted above, subjects with other invasive malignancies, who had any evidence of the other cancer present within the last 3 years or whose previous cancer treatment contraindicates this protocol therapy, are excluded
* Known acute hepatitis
* acute infectious disease with need for intravenous antibiosis
* immunodeficiency
* Active coronaryarterial disease: Myocardinfarct or instable Angina pectoris within 6 months before study inclusion: coronary artery disease in anamnesis can be included, assumed a normal stress-electrocardiogram finding within 30 days before study inclusion
* Cardiac insufficiency NYHA ≥2 classif. of New York Heart Association
* Hypertension ≥140/90 mm Hg
* Poorly controlled cardiac arrythmia despite medication (patients with frequencey-controlled atrial fibrillation can participate)
* Peripheral vascular disease ≥grade 3 (e.g. symptomatic and affecting activities of everyday-life, intervention or revision necessary)
* Renal insufficiency Serumcreatininvalues ≥1,5 times the ULN or GFR <60ml/min
* Cerebrovascular disease in anamnesis
* Patients with another severe medical problem-independent of cancer-which excludes study participation
* Known allergies to Carboplatin or Cisplatin
* extended intraperitoneal adhesions at time of secondary cytoreductive operation, which makes administration of intraperitioneal chemotherapy impossible
* Life expectancy <12 weeks

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Elevation of side-effects and postoperative complication-rate | 24 months
  Observation, classification and graduation of side-effects through NCI Common Terminology Criteria for Adverse Events version 4.03 ["safety issue"]

SECONDARY OUTCOMES:
Survey of quality of life per EORTC evaluated questionnaires | 24 months
  Using EORTC -QLQ-C30 and EORTC QLQ-OV28, at study initiation, postoperative, before systemic chemotherapy and afterwards
Recording of PFS (progession free survival) | 24 months
  Recording of PFS (progession free survival) of the patients in a time-span of 24 months [kein "safety issue"]

CONTACTS AND LOCATIONS:
Overall Officials: Lukas Hefler, Prim. Dr., Principal Investigator — Krankenhaus der Barmherzigen Schwestern Linz
Locations (1):
- Department of gynaecology, Ordensklinikum Linz Ges.m.b.H, Barmherzige Schwestern, Linz, Austria